CLINICAL TRIAL: NCT07339137
Title: The Effects of Platelet-rich Plasma (PRP) Injections Administered Into Intra-articular and Periarticular Regions Under Ultrasound Guidance in Chronic Knee Osteoarthritis on Pain, Function, Activities of Daily Living, Medial Collateral Ligament (MCL) and Distal Femoral Cartilage Thickness
Brief Title: The Effects of Intra-articular and Peri-articular Platelet-rich Plasma (PRP) Injections ın Chronic Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, RIDVAN ÇELİK, Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-25-9883
Record Dates: First submitted 2026-01-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Platelet Rich Plasma Injection; Ultrasonography; Gonarthrosis
Keywords: knee osteoarthritis; periarticular; PRP; USG; Femoral Cartilage; Medial Collateral Ligament
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: This randomized, parallel-group study will compare the effects of conservative treatment alone, intra-articular platelet-rich plasma (PRP) injections in addition to conservative treatment, and combined intra-articular and peri-articular PRP injections in patients with chronic knee osteoarthritis (OA). Participants will be assigned to one of three intervention groups. Clinical and ultrasonographic outcomes will be assessed at baseline, 1 week after completion of treatment, and 3 months after completion of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Patients receiving guidance on conservative exercise therapy and lifestyle chang
  Interventions: Behavioral: Conservative Therapy
- Intra-articular PRP (Active Comparator): Patients receiving intra-articular PRP therapy in addition to guidance on conservative exercise therapy and lifestyle chang
  Interventions: Behavioral: Conservative Therapy; Procedure: Intra-Articular PRP
- Combinated PRP (Intra and peri-articular PRP) (Active Comparator): Patients receiving combined (periarticular and intraarticular PRP therapy) in addition to guidance on conservative exercise therapy and lifestyle chang
  Interventions: Behavioral: Conservative Therapy; Procedure: Intra-Articular PRP; Procedure: Peri-Articular PRP

INTERVENTIONS:
Behavioral: Conservative Therapy — Patients will receive guidance on conservative exercise therapy and lifestyle modifications. Exercise instruction forms will be provided, and patients will be shown how to perform the exercises correctly. Strengthening, stretching, and joint range of motion exercises targeting the quadriceps and hamstring muscle groups will be performed twice daily for 10 repetitions throughout the treatment period. Adherence will be monitored during follow-up visits.
Procedure: Intra-Articular PRP — Patients will receive intra-articular platelet-rich plasma (PRP) injections three times at one-week intervals. Following the PRP injections, patients will receive standard post-procedure recommendations, including resting the knee joint for 1-2 days, avoiding aggressive exercise, refraining from using nonsteroidal anti-inflammatory drugs (NSAIDs), and applying warm compresses as needed.
  Arms: Combinated PRP (Intra and peri-articular PRP); Intra-articular PRP
Procedure: Peri-Articular PRP — Patients will receive peri-articular platelet-rich plasma (PRP) injections three times at one-week intervals. Following the PRP injections, patients will receive standard post-procedure recommendations, including resting the knee joint for 1-2 days, avoiding aggressive exercise, refraining from using nonsteroidal anti-inflammatory drugs (NSAIDs), and applying warm compresses as needed.
  Peri-articular injections will be administered under ultrasound (USG) guidance to the origin and insertion sites of the medial collateral ligament (MCL), relevant joint areas, and the insertion points of the pes anserinus tendons.
  Arms: Combinated PRP (Intra and peri-articular PRP)

SUMMARY:
The primary objective of this study is to evaluate and compare the effectiveness of ultrasound-guided combined intra-articular and peri-articular platelet-rich plasma (PRP) injections with intra-articular PRP injections alone in patients with chronic knee osteoarthritis (OA). The study specifically examines the effects of these treatment approaches on pain, physical function, activities of daily living, and structural parameters, including medial collateral ligament (MCL) thickness and distal femoral cartilage thickness.

Osteoarthritis is a degenerative joint disease characterized by progressive cartilage erosion, osteophyte formation, and subchondral sclerosis, leading to pain, stiffness, and functional disability. It is the most common form of arthritis and a leading cause of disability worldwide, affecting approximately 300 million individuals. Although the knee is the most frequently involved joint, OA is now recognized as a whole-joint disease, involving not only cartilage degeneration but also pathological changes in subchondral bone, synovium, and surrounding extra-articular structures.

Platelet-rich plasma is an autologous concentration of platelets suspended in a small volume of plasma and contains a variety of bioactive growth factors, such as transforming growth factor-beta (TGF-β), platelet-derived growth factor (PDGF), and vascular endothelial growth factor (VEGF). These factors play a crucial role in promoting cell proliferation, angiogenesis, and tissue repair. In knee OA, PRP has been shown to reduce matrix metalloproteinase (MMP) activity, particularly MMP-13, enhance endogenous hyaluronic acid production, and support chondrogenesis. Although intra-articular PRP injections are widely accepted as a safe and effective treatment and have demonstrated superiority over placebo and hyaluronic acid in long-term follow-up studies, most existing research has focused exclusively on intra-articular applications.

Knee OA is a multifactorial condition frequently associated with extra-articular pathologies, including ligament laxity, peri-articular edema, and soft tissue inflammation. Limiting treatment to the intra-articular space alone may therefore overlook these important contributors to pain and functional impairment. Emerging evidence suggests that a combined treatment approach targeting both intra-articular and peri-articular structures may provide superior outcomes in terms of pain reduction and functional improvement.

This prospective randomized controlled trial will include 42 patients aged 40-65 years with chronic knee OA classified as Kellgren-Lawrence grade 2 or 3. Participants will be randomly assigned to one of three groups: a control group receiving conservative treatment only (exercise therapy and lifestyle modifications), a group receiving conservative treatment plus ultrasound-guided intra-articular PRP injections, and a third group receiving conservative treatment plus combined ultrasound-guided intra-articular and peri-articular PRP injections targeting the MCL and pes anserinus regions.

Clinical outcomes will be assessed using validated instruments, including the Visual Analog Scale (VAS), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Short Form-36 (SF-36) Quality of Life Scale. In addition, ultrasonographic measurements of MCL thickness and distal femoral cartilage thickness will be performed to evaluate structural changes. By investigating the additional value of peri-articular PRP injections, this study aims to contribute to the development of more comprehensive and effective injection protocols for the management of chronic knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a dynamic condition characterized by a disruption in the balance between anabolic and catabolic processes of joint matrix molecules, favoring catabolism. Although OA is primarily recognized for cartilage degeneration, its pathogenesis involves a complex inflammatory and degenerative process affecting the entire joint unit, including subchondral bone, synovium, and surrounding soft tissues. Platelet-rich plasma (PRP) has emerged as an effective and safe treatment option for knee OA, particularly for patients who are unable to tolerate oral pharmacological therapies or wish to delay surgical intervention. PRP promotes tissue healing through the release of various growth factors from platelet alpha granules, which enhance cellular proliferation, stimulate angiogenesis, and reduce the activity of inflammatory mediators.

Current literature predominantly focuses on the efficacy of intra-articular PRP applications. However, knee OA is a multifactorial disease frequently accompanied by extra-articular pathologies, such as ligament laxity, edema, and peri-articular soft tissue inflammation. An exclusive focus on the intra-articular space may therefore overlook these extra-articular contributors to pain and functional impairment. This study is based on the hypothesis that a combined treatment approach targeting both the intra-articular environment and peri-articular structures-specifically the medial collateral ligament (MCL) and pes anserinus-will result in superior clinical outcomes compared to intra-articular treatment alone.

The use of ultrasound (USG) guidance in this study ensures accurate needle placement and enables objective assessment of structural changes. While intra-articular PRP has been shown to be more effective than hyaluronic acid or saline injections at 6- to 12-month follow-ups, evidence regarding the additional benefits of peri-articular PRP injections remains limited. To our knowledge, this study will be among the few randomized controlled trials comparing combined intra-articular and peri-articular PRP application with isolated intra-articular PRP treatment. Moreover, by evaluating changes in MCL thickness and distal femoral cartilage thickness using USG, this study aims to provide objective structural data to the existing literature.

In this prospective randomized controlled trial, 42 patients will be allocated into three groups. Group 1 (control group) will receive conservative treatment consisting of exercise therapy, lifestyle modifications, and patient education. Group 2 will receive conservative treatment in addition to three sessions of USG-guided intra-articular PRP injections administered at one-week intervals. Group 3 will receive conservative treatment plus three sessions of combined USG-guided intra-articular and peri-articular PRP injections, with peri-articular injections targeting the MCL origin and insertion sites as well as the pes anserinus tendon insertion.

All PRP applications will be performed using a standardized preparation kit and a photo-activation system to maximize growth factor release. Patients will be evaluated at baseline and followed up at 1 week and 3 months post-treatment using validated outcome measures, including the Visual Analog Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and Short Form-36 (SF-36), along with ultrasonographic assessments to evaluate pain, function, and structural regeneration.

ELIGIBILITY:
Inclusion Criteria

* Age between 40 and 65 years.
* Patients with significant medial knee pain who have not responded to conservative treatment for at least 3 months.
* Patients diagnosed with knee osteoarthritis according to the American College of Rheumatology (ACR) criteria and with Kellgren-Lawrence grade 2 or 3 radiographic osteoarthritis.
* Intact cognitive function.
* Willingness to participate in the study and provide signed informed consent.
* Visual Analog Scale (VAS) score of 4 or higher.

Exclusion Criteria

* History of previous knee trauma or surgery.
* Physical therapy, intra-articular steroid, or hyaluronic acid injections in the knee within the last 3 months.
* Active oncological diseases.
* Local infection, sepsis, wounds, or scars in the injection area.
* Systemic infections, hepatitis, or immunosuppression.
* Bleeding diathesis or irregular International Normalized Ratio (INR) due to oral warfarin use.
* Inflammatory arthropathies.
* Uncontrolled hypertension, uncontrolled diabetes mellitus, decompensated heart failure, coronary artery disease, or asthma.
* Suspected or confirmed pregnancy.
* Use of corticosteroids or opioids.
* Anemia.
* Body mass index (BMI) greater than 35.
* Allergy to citrate.
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within the last week that may affect platelet function analyzer-100 (PFA-100) activity.
* Physical examination findings suggestive of patellar retinaculum, meniscus, or cruciate ligament injury.
* General health impairment or lack of cooperation.
* Refusal to participate in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale) | Pain measurements using the VAS will be obtained at baseline (week 0), 1 week after completion of treatment (week 3), and 3 months after completion of treatment (week 14).
  The visual analog scale (VAS) is a widely accepted measurement tool in the scientific literature used to quantify subjective variables that cannot be directly measured numerically. It consists of a 100-mm horizontal line, with each end representing the extreme limits of the parameter being assessed, ranging from no pain to very severe pain. Patients are asked to mark the point on the line that best reflects their current pain intensity. The distance measured from the no-pain endpoint to the patient's mark indicates the level of pain. The VAS is a safe, easy-to-use, and valid instrument for assessing pain intensity.
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | The WOMAC will be assessed at baseline (week 0), 1 week after completion of treatment (week 3), and 3 months after completion of treatment (week 14).
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a valid and reliable disease-specific instrument widely used to assess disability in patients with osteoarthritis. It consists of three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Each item is scored on a Likert scale ranging from 0 to 4, reflecting the level of impairment. Subscale scores are calculated separately and combined to yield a total score ranging from 0 to 100, with higher scores indicating increased pain and stiffness and greater impairment in physical function. The Turkish validity and reliability of the WOMAC were established by Tüzün and colleagues.

SECONDARY OUTCOMES:
SF-36 (Short Form 36 Health Survey) | Quality of life will be assessed using the SF-36 at baseline (week 0), 1 week after completion of treatment (week 3), and 3 months after completion of treatment (week 14).
  The Short Form-36 (SF-36) is a widely used instrument for assessing patients' overall health status and quality of life, with established validity and reliability in Turkish populations. The scale consists of 36 items across 8 subscales: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional health, and mental health. Each item is scored individually, and scores are calculated to produce a total score ranging from 0 to 100, with higher scores indicating better quality of life and lower scores indicating poorer quality of life.
Distal femoral cartilage thickness | Distal femoral cartilage thickness will be measured at baseline (week 0), 1 week after completion of treatment (week 3), and 3 months after completion of treatment (week 14) for each participant.
  The distal femoral cartilage thickness of all participants will be assessed by the same researcher experienced in musculoskeletal ultrasonography using an ultrasound device (Logiq P5, GE Medical Systems, USA) equipped with a linear probe operating at a frequency of 5-12 megahertz (MHz). Measurements will be performed with participants in the supine position and knees in maximum flexion. The ultrasound probe will be positioned perpendicular to the articular surface of the femur by placing it transversely on the upper edge of the patella. Cartilage will be identified as a hypoechoic structure located between the suprapatellar fat pad and the bone cortex. Thickness measurements will be taken at three sites: the midpoint of the medial condyle, the intercondylar notch, and the lateral condyle. Measurements will be based on the distance between the bone-cartilage interface and the cartilage-fat pad interface.
Medial Collateral Ligament thickness | Medial collateral ligament (MCL) thickness will be measured at baseline (week 0), 1 week after completion of treatment (week 3), and 3 months after completion of treatment (week 14) for each participant.
  The medial collateral ligament (MCL) of all participants will be assessed by the same researcher experienced in musculoskeletal ultrasonography using a linear probe ultrasound device (Logiq P5, GE Medical Systems, USA) operating at a frequency of 5-12 megahertz (MHz). During assessment, participants will be positioned supine with their knees fully extended. After visualizing the joint space, the MCL will be imaged in the vertical plane along the medial side of the knee. Thickness measurements will be taken at two points: approximately 1 cm proximal to the joint line on the femoral side and 1 cm distal to the joint line on the tibial side.

CONTACTS AND LOCATIONS:
Overall Officials: Emre ADIGÜZEL, Prof. Dr., Study Director — Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital
Locations (1):
- Ankara Bilkent City Hospital, Physical Therapy and Rehabilitation Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen L, Yuan T, Chen S, Xie X, Zhang C. The temporal effect of platelet-rich plasma on pain and physical function in the treatment of knee osteoarthritis: systematic review and meta-analysis of randomized controlled trials. J Orthop Surg Res. 2017 Jan 23;12(1):16. doi: 10.1186/s13018-017-0521-3. PMID 28115016
- [Background] Sit RWS, Wu RWK, Law SW, Zhang DD, Yip BHK, Ip AKK, Rabago D, Reeves KD, Wong SYS. Intra-articular and extra-articular platelet-rich plasma injections for knee osteoarthritis: A 26-week, single-arm, pilot feasibility study. Knee. 2019 Oct;26(5):1032-1040. doi: 10.1016/j.knee.2019.06.018. Epub 2019 Jul 30. PMID 31375446
- [Background] Tao X, Aw AAL, Leeu JJ, Bin Abd Razak HR. Three Doses of Platelet-Rich Plasma Therapy Are More Effective Than One Dose of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Systematic Review and Meta-analysis. Arthroscopy. 2023 Dec;39(12):2568-2576.e2. doi: 10.1016/j.arthro.2023.05.018. Epub 2023 May 24. PMID 37236291
- [Background] Mascarenhas R, Saltzman BM, Fortier LA, Cole BJ. Role of platelet-rich plasma in articular cartilage injury and disease. J Knee Surg. 2015 Feb;28(1):3-10. doi: 10.1055/s-0034-1384672. Epub 2014 Jul 28. PMID 25068847
- [Background] Aras B, Celik R, Tezen O, Adiguzel E. Associations of medial collateral ligament and cartilage thickness with clinical outcomes in medial knee osteoarthritis: a cross-sectional study. Clin Rheumatol. 2026 Jan;45(1):441-447. doi: 10.1007/s10067-025-07809-x. Epub 2025 Nov 17. PMID 41247668
- [Background] Pane RV, Setiyaningsih R, Widodo G, Al Hajiri AZZ, Salsabil JR. Femoral Cartilage Thickness in Knee Osteoarthritis Patients and Healthy Adults: An Ultrasound Measurement Comparison. ScientificWorldJournal. 2023 Feb 17;2023:3942802. doi: 10.1155/2023/3942802. eCollection 2023. PMID 36845755
- [Background] Testa G, Giardina SMC, Culmone A, Vescio A, Turchetta M, Cannavo S, Pavone V. Intra-Articular Injections in Knee Osteoarthritis: A Review of Literature. J Funct Morphol Kinesiol. 2021 Feb 3;6(1):15. doi: 10.3390/jfmk6010015. PMID 33546408